CLINICAL TRIAL: NCT06118450
Title: A Prospective, Multi-center Clinical Trial for Evaluating the Effectiveness and Safety of Online Coronary Angiography-Derived Index of Microcirculatory Resistance in STEMI Patients (Flash IV)
Brief Title: Clinical Trial for Evaluating the Effectiveness and Safety of Online caIMR in STEMI Patients
Acronym: FlashIV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Collaborators: RainMed Medical Group (Industry)
Responsible Party: Sponsor
Other Study IDs: XYFY2023-QL152-02
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Microvascular Coronary Artery Disease; STEMI
Keywords: STEMI; caIMR; coronary microvascular disease
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Microvascular Angina

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high caIMR: caIMR≥25
  Interventions: Other: Non-intervention
- low caIMR: caIMR<25
  Interventions: Other: Non-intervention

INTERVENTIONS:
Other: Non-intervention — non-intervention

SUMMARY:
Despite the success of restoration of epicardial blood flow by the primary percutaneous coronary intervention (PPCI), approximately a half of patients with ST-segment elevation myocardial infarction (STEMI) have failed myocardial reperfusion, as reflected by microvascular obstruction (MVO) and intramyocardial haemorrhage (IMH). The coronary angiography-derived index of microvascular resistance (caIMR) is a brand new method for assessing coronary microcirculation in ischemia and no obstructive coronary artery disease (INOCA). In this trial, the investigators aim to verify the safety and effectiveness of caIMR in STEMI who underwent primary PCI. The investigators will immediately measure the caIMR of patients who successfully underwent pPCI, and combine the caIMR with the long-term prognosis, to verify the prognostic performance of caIMR.

DETAILED DESCRIPTION:
Despite the success of restoration of epicardial blood flow by the primary percutaneous coronary intervention (PPCI), approximately a half of patients with ST-segment elevation myocardial infarction (STEMI) have failed myocardial reperfusion, as reflected by microvascular obstruction (MVO) and intramyocardial haemorrhage (IMH). There are many defects in the current measurement technology, such as non-timely, long measurement time, high price, potential risk of gadolinium contrast agent.

The index of microcirculatory resistance (IMR) is a readily available, wire-based approach for assessing microvascular dysfunction immediately post-stenting for STEMI. The parameter has been used to characterize MVO, was associated with infarct size, and subsequent cardiac death and heart failure. However, the application of IMR in clinical practice remains limited, primarily due to the requirement of a pressure-temperature sensor wire and hyperaemic agents, which add complexity and time.

The development of functional coronary angiography has enabled the estimation of IMR based on angiography alone. The coronary angiography-derived index of microvascular resistance (caIMR) has shown good diagnostic accuracy compared with wire-based invasive IMR. This simple alternative index showed an association with extent of MVO and was of prognostic importance. In this trial, the investigators aim to verify the safety and effectiveness of caIMR in STEMI who underwent primary PCI. The investigators will immediately measure the caIMR of patients who successfully underwent pPCI, and combine the caIMR with the long-term prognosis, to verify the prognostic performance of caIMR.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 80, regardless of gender;
* Initially diagnosed as STEMI and underwent primary PCI;
* Voluntarily participated in this trial and signed the informed consent form.

Exclusion Criteria:

* Coronary angiography shows that PCI is not suitable;
* Past history of coronary artery bypass grafting (CABG);
* Past history of heart failure;
* Past history of myocardial infarction;
* Primary or secondary cardiomyopathy or heart valve disease;
* Patients with renal insufficiency (eGFR<30ml/min (1.73m^2)) or patients undergoing dialysis;
* Cardiogenic shock
* Persistent left or right coronary ostium lesion after target vessel PCI;
* Immediate effect of target vessel PCI is unsatisfactory [such as thrombolysis in myocardial infarction (TIMI) flow < grade 2, dissection that restricted blood flow, side branch occlusion (diameter>1.5mm), exist distal embolism or angiographically visible thrombus];
* Target vessel exist coronary fistula or myocardial bridge (lumen constriction >50%);
* The target vessel cannot clearly expose the lesion in two positions with an included angle ≥ 30 degrees;
* Severe systemic infection
* Patients with malignant wasting disease, with an estimated survival of less than 1 year;
* The subject is participating in another clinical researches, and the primary endpoint has not been reached;
* The investigator believes that the subject has other conditions that are not suitable for clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aged between 18 and 80, regardless of gender. Initially diagnosed as STEMI and underwent primary PCI.
Sampling Method: Probability Sample
Enrollment: 335 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE ) | 12 months
  Rate of MACE. MACE was defined as a composite endpoint of cardiac death, myocardial reinfarction, readmission for heart failure, and unplanned readmission for ischemia.

SECONDARY OUTCOMES:
MACE | 1 month; 6months
  Rate of MACE. MACE was defined as a composite outcome of cardiac death, myocardial reinfarction, readmission for heart failure, and unplanned readmission for ischemia.
Outcome events for each category | 12 months
  Rate of cardiac death, rate of myocardial reinfarction, rate of readmission for heart failure, and rate of unplanned readmission for ischemia.
Stroke | 12 months
  incidence rate
Malignant arrhythmia | 12 months
  incidence rate
Target vessel failure (TVF) | 12 months
  Rate of TVF. TVF was defined as a combined outcome, consisting of revascularization, infarction and death for target vessel

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Beijing Luhe Hospital.Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - The First People'S Hospital of Lianyungang, Lianyungang, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - General Hospital of Xuzhou Mining Group, Xuzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Xuzhou First People's Hospital, Xuzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li J, Gong Y, Wang W, Yang Q, Liu B, Lu Y, Xu Y, Huo Y, Yi T, Liu J, Li Y, Xu S, Zhao L, Ali ZA, Huo Y. Accuracy of computational pressure-fluid dynamics applied to coronary angiography to derive fractional flow reserve: FLASH FFR. Cardiovasc Res. 2020 Jun 1;116(7):1349-1356. doi: 10.1093/cvr/cvz289. PMID 31693092
- [Background] Zhang D, Lv S, Song X, Yuan F, Xu F, Zhang M, Yan S, Cao X. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention: a meta-analysis. Heart. 2015 Mar;101(6):455-62. doi: 10.1136/heartjnl-2014-306578. Epub 2015 Jan 30. PMID 25637372
- [Background] Davies JE, Sen S, Dehbi HM, Al-Lamee R, Petraco R, Nijjer SS, Bhindi R, Lehman SJ, Walters D, Sapontis J, Janssens L, Vrints CJ, Khashaba A, Laine M, Van Belle E, Krackhardt F, Bojara W, Going O, Harle T, Indolfi C, Niccoli G, Ribichini F, Tanaka N, Yokoi H, Takashima H, Kikuta Y, Erglis A, Vinhas H, Canas Silva P, Baptista SB, Alghamdi A, Hellig F, Koo BK, Nam CW, Shin ES, Doh JH, Brugaletta S, Alegria-Barrero E, Meuwissen M, Piek JJ, van Royen N, Sezer M, Di Mario C, Gerber RT, Malik IS, Sharp ASP, Talwar S, Tang K, Samady H, Altman J, Seto AH, Singh J, Jeremias A, Matsuo H, Kharbanda RK, Patel MR, Serruys P, Escaned J. Use of the Instantaneous Wave-free Ratio or Fractional Flow Reserve in PCI. N Engl J Med. 2017 May 11;376(19):1824-1834. doi: 10.1056/NEJMoa1700445. Epub 2017 Mar 18. PMID 28317458
- [Background] Lerman A, Holmes DR, Herrmann J, Gersh BJ. Microcirculatory dysfunction in ST-elevation myocardial infarction: cause, consequence, or both? Eur Heart J. 2007 Apr;28(7):788-97. doi: 10.1093/eurheartj/ehl501. Epub 2007 Mar 8. PMID 17347176
- [Background] Bolognese L, Carrabba N, Parodi G, Santoro GM, Buonamici P, Cerisano G, Antoniucci D. Impact of microvascular dysfunction on left ventricular remodeling and long-term clinical outcome after primary coronary angioplasty for acute myocardial infarction. Circulation. 2004 Mar 9;109(9):1121-6. doi: 10.1161/01.CIR.0000118496.44135.A7. Epub 2004 Feb 16. PMID 14967718
- [Background] Hombach V, Grebe O, Merkle N, Waldenmaier S, Hoher M, Kochs M, Wohrle J, Kestler HA. Sequelae of acute myocardial infarction regarding cardiac structure and function and their prognostic significance as assessed by magnetic resonance imaging. Eur Heart J. 2005 Mar;26(6):549-57. doi: 10.1093/eurheartj/ehi147. Epub 2005 Feb 15. PMID 15713695
- [Background] Wu KC, Zerhouni EA, Judd RM, Lugo-Olivieri CH, Barouch LA, Schulman SP, Blumenthal RS, Lima JA. Prognostic significance of microvascular obstruction by magnetic resonance imaging in patients with acute myocardial infarction. Circulation. 1998 Mar 3;97(8):765-72. doi: 10.1161/01.cir.97.8.765. PMID 9498540
- [Background] Eitel I, de Waha S, Wohrle J, Fuernau G, Lurz P, Pauschinger M, Desch S, Schuler G, Thiele H. Comprehensive prognosis assessment by CMR imaging after ST-segment elevation myocardial infarction. J Am Coll Cardiol. 2014 Sep 23;64(12):1217-26. doi: 10.1016/j.jacc.2014.06.1194. PMID 25236513
- [Background] Cuculi F, De Maria GL, Meier P, Dall'Armellina E, de Caterina AR, Channon KM, Prendergast BD, Choudhury RP, Forfar JC, Kharbanda RK, Banning AP. Impact of microvascular obstruction on the assessment of coronary flow reserve, index of microcirculatory resistance, and fractional flow reserve after ST-segment elevation myocardial infarction. J Am Coll Cardiol. 2014 Nov 4;64(18):1894-904. doi: 10.1016/j.jacc.2014.07.987. Epub 2014 Oct 27. PMID 25444143
- [Background] De Maria GL, Alkhalil M, Wolfrum M, Fahrni G, Borlotti A, Gaughran L, Dawkins S, Langrish JP, Lucking AJ, Choudhury RP, Porto I, Crea F, Dall'Armellina E, Channon KM, Kharbanda RK, Banning AP. Index of Microcirculatory Resistance as a Tool to Characterize Microvascular Obstruction and to Predict Infarct Size Regression in Patients With STEMI Undergoing Primary PCI. JACC Cardiovasc Imaging. 2019 May;12(5):837-848. doi: 10.1016/j.jcmg.2018.02.018. Epub 2018 Apr 18. PMID 29680355
- [Background] Fahrni G, Wolfrum M, De Maria GL, Cuculi F, Dawkins S, Alkhalil M, Patel N, Forfar JC, Prendergast BD, Choudhury RP, Channon KM, Banning AP, Kharbanda RK. Index of Microcirculatory Resistance at the Time of Primary Percutaneous Coronary Intervention Predicts Early Cardiac Complications: Insights From the OxAMI (Oxford Study in Acute Myocardial Infarction) Cohort. J Am Heart Assoc. 2017 Nov 7;6(11):e005409. doi: 10.1161/JAHA.116.005409. PMID 29113999
- [Background] Fearon WF, Low AF, Yong AS, McGeoch R, Berry C, Shah MG, Ho MY, Kim HS, Loh JP, Oldroyd KG. Prognostic value of the Index of Microcirculatory Resistance measured after primary percutaneous coronary intervention. Circulation. 2013 Jun 18;127(24):2436-41. doi: 10.1161/CIRCULATIONAHA.112.000298. Epub 2013 May 16. PMID 23681066
- [Background] Fearon WF, Shah M, Ng M, Brinton T, Wilson A, Tremmel JA, Schnittger I, Lee DP, Vagelos RH, Fitzgerald PJ, Yock PG, Yeung AC. Predictive value of the index of microcirculatory resistance in patients with ST-segment elevation myocardial infarction. J Am Coll Cardiol. 2008 Feb 5;51(5):560-5. doi: 10.1016/j.jacc.2007.08.062. PMID 18237685
- [Background] McGeoch R, Watkins S, Berry C, Steedman T, Davie A, Byrne J, Hillis S, Lindsay M, Robb S, Dargie H, Oldroyd K. The index of microcirculatory resistance measured acutely predicts the extent and severity of myocardial infarction in patients with ST-segment elevation myocardial infarction. JACC Cardiovasc Interv. 2010 Jul;3(7):715-22. doi: 10.1016/j.jcin.2010.04.009. PMID 20650433
- [Background] Ai H, Feng Y, Gong Y, Zheng B, Jin Q, Zhang HP, Sun F, Li J, Chen Y, Huo Y, Huo Y. Coronary Angiography-Derived Index of Microvascular Resistance. Front Physiol. 2020 Dec 16;11:605356. doi: 10.3389/fphys.2020.605356. eCollection 2020. PMID 33391020
- [Background] Abdu FA, Liu L, Mohammed AQ, Yin G, Xu B, Zhang W, Xu S, Lv X, Fan R, Feng C, Shi T, Huo Y, Xu Y, Che W. Prognostic impact of coronary microvascular dysfunction in patients with myocardial infarction with non-obstructive coronary arteries. Eur J Intern Med. 2021 Oct;92:79-85. doi: 10.1016/j.ejim.2021.05.027. Epub 2021 Jun 4. PMID 34092485
- [Background] Choi KH, Dai N, Li Y, Kim J, Shin D, Lee SH, Joh HS, Kim HK, Jeon KH, Ha SJ, Kim SM, Jang MJ, Park TK, Yang JH, Song YB, Hahn JY, Doh JH, Shin ES, Choi SH, Gwon HC, Lee JM. Functional Coronary Angiography-Derived Index of Microcirculatory Resistance in Patients With ST-Segment Elevation Myocardial Infarction. JACC Cardiovasc Interv. 2021 Aug 9;14(15):1670-1684. doi: 10.1016/j.jcin.2021.05.027. PMID 34353599
- [Background] Duan Y, Wang Y, Zhang M, Li Z, Chen L, Miao H, Pei S, Lu Y, Wang Z. Computational Pressure-Fluid Dynamics Applied to Index of Microcirculatory Resistance, Predicting the Prognosis of Drug-Coated Balloons Compared With Drug-Eluting Stents in STEMI Patients. Front Physiol. 2022 May 24;13:898659. doi: 10.3389/fphys.2022.898659. eCollection 2022. PMID 35685283